CLINICAL TRIAL: NCT05082077
Title: Global Utilization and Registry Database for Improved Preservation of Donor Livers
Status: Enrolling by invitation | Type: Observational
Sponsor: Paragonix Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: PGX-005
Record Dates: First submitted 2021-09-24; First posted 2021-10-18 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-07

CONDITIONS: Liver Diseases; Liver Dysfunction; Liver Transplant Disorder; Liver Transplant Rejection
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- LIVERguard patient: Patients whose donor liver was transported with the LiverGuard device.
  Interventions: Device: LIVERguard
- Standard Transport Patients: Patients whose donor liver was transported with a method other than the LiverGuard

INTERVENTIONS:
Device: LIVERguard — The LIVERguard is an FDA cleared and is a CE-marked medical device intended to be used for the static hypothermic preservation of livers during transportation and eventual transplantation into a recipient using cold storage solutions indicated for use with the liver. The intended organ storage time for the LIVERguard is up to 16 hours.
  Groups: LIVERguard patient

SUMMARY:
The objective of this registry is to collect and evaluate various clinical effectiveness parameters in patients with transplanted donor liver that were preserved and transported within the LIVERguard system, as well as retrospective standard of care patients

DETAILED DESCRIPTION:
GUARDIAN-Liver is a post-market, observational registry of adult and pediatric liver transplant recipient patients whose donor liver was preserved and transported within the LIVERguard. The data is being collected retrospectively from medical records of patients already transplanted before the initiation of the registry and any new patients who meet the eligibility criteria.

About 1000 male and female subjects meeting the study inclusion and exclusion criteria will be enrolled into the study at about 20 clinical sites.

Candidates that fit the eligibility criteria and have had their donor liver transported with a Paragonix product or a standard of care method can be enrolled. The baseline characteristics and outcomes of the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Donor and donor liver matched to the recipient based upon institutional medical practice
* Registered male or female primary liver transplant candidates

Exclusion Criteria:

* Donor and donor liver that do not meet institutional clinical requirements for transplantation
* Living donors
* Pediatric recipients (under 18)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received a liver transplant at centers that use the LIVERguard device
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Graft Failure | Post-transplant through 1 year post
  The percentage of subjects in each cohort who develop graft failure post-transplant
Early allograft dysfunction | 7 days post transplant
  The percentage of subjects in each cohort who early allograft failure post-transplant
Rejection | Post-transplant through 1 year post
  The percentage of subjects in each cohort who experience rejection post-transplant
Primary Non-function | Post transplant to 7 days post-transplant
  The percentage of subjects in each cohort who experience primary non-function post-transplant
Survival | Transplant through 1 year post-transplant
  The percentage of subjects in each cohort who survive through 1 year post-transplant
Length of Stay | 1 year
  How many days the patient stays in the hospital post-transplant
Length of ICU stay | 1 year
  How many days the patient stayed in the ICU post-transplant

SECONDARY OUTCOMES:
Hospitalizations | post-transplant through 1 year
  Amount of times patient is rehospitalized after discharge post-transplant
Biliary complications | post-transplant through 1 year post-transplant
  Percentage of patients that experience biliary strictures in each cohort as determined by lab work

CONTACTS AND LOCATIONS:
Overall Officials: Jason Vanatta, MD, Principal Investigator — Methodist Le Bonheur Healthcare
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Stanford, California
  - University of Florida, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of Nebraska, Omaha, Nebraska
  - Duke University, Durham, North Carolina
  - University of Washington, Seattle, Washington